CLINICAL TRIAL: NCT06557434
Title: AV-23-001 AVAVA MIRIA Pilot Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AVAVA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-23-001
Record Dates: First submitted 2023-12-11; First posted 2024-08-16 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Wrinkle; Acne Scars - Mixed Atrophic and Hypertrophic; Pigmented Lesions; Skin Laxity; Scars
Keywords: MIRIA; Laser; Wrinkles; Acne Scars; Skin Laxity; Skin Improvement; non-ablative
MeSH Terms: conditions — Hypertrophy; Cutis Laxa; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treated Cohort (Experimental): Experimental: Treatment with the MIRIA Laser 3-4 experimental treatments at 4-6 week intervals. Refine usage of device
  Interventions: Device: MIRIA

INTERVENTIONS:
Device: MIRIA — The MIRIA Skin Treatment System is a 1550nm-based laser system indicated for use in dermatologic procedures requiring the coagulation of soft tissue, as well as for skin resurfacing procedures.

SUMMARY:
This non-significant risk study is intended to demonstrate the use of the MIRIA Skin Treatment System can show improvement in dermatologic conditions currently indicated for treatment with a laser (such as, but not limited to, benign pigmented lesions, benign cutaneous lesions, wrinkles, textural irregularities, or scars). The study is also intended to assist in determination of the optimal laser configuration and treatment parameters that most consistently yield results.

DETAILED DESCRIPTION:
This study is intended to allow clinical evaluation of the feasibility of the MIRIA Skin Treatment System, referred to herein as the SR Skin Rejuvenation Laser, for the treatment of dermatologic conditions currently indicated for treatment with a laser (such as, but not limited to, benign pigmented lesions, benign cutaneous lesions, wrinkles, textural irregularities, or scars). This clinical evaluation is being performed under an investigational protocol to formally collect data for the treatment of different dermatologic conditions.

This prospective, non-randomized, controlled study will include subjects with dermatologic conditions that are currently indicated for treatment with a laser who are willing to have sites exposed to the MIRIA Laser and who agree to comply with the study requirements during the follow-up period, a minimum of 3 months and a maximum of 18 months. Some areas with the dermatologic condition may be left as a control for the treated section. Subjects may also be directed to use some topical cream or lotion for up to 1 month prior to the laser procedure or during the duration of the study, according to the Investigator's standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Dermatologic condition currently indicated for laser treatment OR the subject is to be enrolled for assessment of treatment parameters on normal skin.
3. Willingness to have multiple areas exposed.
4. Willingness to have digital photographs taken of treatment area(s) and agreement with use of photographs for presentation, educational, or marketing purposes.
5. Willingness to comply with the following during the study, including the follow-up period:

   1. maintain consistent skin care regimen on treated areas.
   2. Willingness to cover treated areas or have very limited sun exposure and, if requested, use an approved sunscreen of SPF 50 or higher.
   3. refrain from using systemic corticosteroids, according to Investigator discretion.
   4. refrain from using topical corticosteroids, retinoids, or prescription skin-lightening medications on the treated areas, according to Investigator discretion.
   5. refrain from any other procedures in the treatment areas.
6. Willingness and ability to comply with study instructions and return for required visits.
7. Subject understands that fees will be collected at the time of treatment ranging from $300 to $3000 per treatment depending upon number of anatomical areas treated. The exact amount will be disclosed and recorded within the consent.
8. Subject has read and signed a written informed consent form.
9. Subject lives within 50 miles of study site.
10. For Males: Willingness to shave facial hair on treatment areas.

    Exclusion Criteria:
11. Skin pathology or condition that could interfere with evaluation of the study procedure, e.g.,
12. Systemic treatment prescribed within previous 6 months (e.g., oral medication such as isotretinoin)
13. Surgical treatment in the target areas within previous 6 months (e.g., laser surgery)
14. Active vitiligo, psoriasis, or eczema in the treatment area
15. The timing of use of fillers, neuromodulators and other cosmetic procedures are at the discretion of the investigator.
16. Topical treatment applied to target areas within the previous 1 month or according to Investigator discretion.
17. Active suntan and unable or unlikely to refrain from tanning within the follow-up period.
18. Artificial tanning in the target areas within the previous 1 month (e.g., spray, lotion, tanning bed) or intention to use artificial tanning within the follow-up period.
19. Active localized or systemic infection, or an open wound in area being treated.
20. Lesions in the treatment areas suspicious for malignancy (skin cancer, melanoma)
21. History of abnormal wound healing or abnormal scarring (e.g., hypertrophic or keloid)
22. History of connective tissue disease, such as lupus or scleroderma.
23. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion (e.g., topicals that produce sensitivity to light may be used in areas other than the target area).
24. History of gold therapy.
25. History of disease stimulated by heat, such as recurrent herpes simplex or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
26. History of radiation to the treatment area or currently undergoing systemic chemotherapy for the treatment of cancer.
27. For Female: Pregnancy or lactation, or intent to become pregnant within the study period.
28. Significant uncontrolled concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
29. History of immunosuppression/immune deficiency disorder or currently using immunosuppressive medications.
30. Current enrollment in a clinical study of any other unapproved investigational drug or device unless it is a noninvasive dermal study for which the subject is in a follow-up period and has other areas of skin that meet the study criteria or has received an investigational drug or been treated with an investigational device within 30 days prior to entering this study.
31. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) | 3 Months
  Scale used to compare before and after images of subjects treated. Scores include the following:
  1. - Very Much Improved
  2. - Much Improved
  3. - Improved
  4. - No Change
  5. - Worse

SECONDARY OUTCOMES:
Subject Questionnaire | Immediate Post Treatment, 3 Months Post Treatment
  Questionnaire that evaluates the subjects impression of the treatment (overall discomfort score, satisfaction with treatment results, notes on treatment sensation).
Adverse Event Assessment | Immediate Post Treatment, 3 Months Post Treatment
  An assessment of side effects and adverse event profile to ensure safety of treatment. Data collected included the event, the duration, the severity, and any other interventions that may occur due to the adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Hyemin Pomerantz, MD, Principal Investigator — AVAVA, Inc.
Locations (2):
- United States (2):
  - Skinfluence Long Island, Dix Hills, New York
  - Laser and Skin Surgery Center of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No